CLINICAL TRIAL: NCT01081847
Title: Malaria Vaccine Phase IB Clinical Trial: Safety and Immunogenicity Study of Plasmodium Vivax CS Derived Synthetic Peptides Formulated in Two Adjuvants
Brief Title: Safety and Immunogenicity Study of Plasmodium Vivax CS Derived Synthetic Peptides Formulated in Two Adjuvants
Acronym: Fase1B
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Malaria Vaccine and Drug Development Center (Other)
Collaborators: Centro médico Imbanaco (Unknown); Asoclinic Inmunología Ltda. (Industry)
Responsible Party: Myriam Arévalo,PhD, Malaria Vaccine and Drug Development Center
Allocation: Randomized | Model: Factorial | Masking: Quadruple
Other Study IDs: MVDC 2003-002; MVDC 2003-002 (Other: MVDC)
Record Dates: First submitted 2010-03-03; First posted 2010-03-05 (Estimated); Last update posted 2010-03-08 (Estimated); Status verified 2010-03

CONDITIONS: Malaria, Vivax
Keywords: Malaria; Synthetic peptides; Plasmodium vivax; Human volunteers
MeSH Terms: conditions — Malaria, Vivax; Malaria | interventions — Peptides; mannide monooleate; montanide ISA 51

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Group A (Active Comparator): Montanide ISA 720 Dose by peptide 50ug
  Interventions: Drug: Peptides (N,R&C) formulated in Montanide ISA 720
- Group B (Active Comparator): Montanide ISA 51 Dose by peptide 50ug
  Interventions: Drug: Peptides (N,R&C) formulated in Montanide ISA 51
- Group C (Active Comparator): Montanide ISA 720 Dose by peptide 100ug
  Interventions: Drug: Peptides (N,R&C) formulated in Montanide ISA 720
- Group D (Active Comparator): Montanide ISA 51 Dose by peptide 100ug
  Interventions: Drug: Peptides (N,R&C) formulated in Montanide ISA 51
- Group E (Placebo Comparator): Control Group. no peptide. Isotonic saline solution
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Peptides (N,R&C) formulated in Montanide ISA 720 — 50 ug
  Other Names: Peptides (N, R & C) from P. vivax CS protein
  Arms: Group A
Drug: Peptides (N,R&C) formulated in Montanide ISA 51 — 50 ug
  Other Names: Peptides (N, R & C) from P. vivax CS protein.
  Arms: Group B
Drug: Peptides (N,R&C) formulated in Montanide ISA 720 — 100 ug
  Other Names: Peptides (N, R & C) from P. vivax CS protein.
  Arms: Group C
Drug: Peptides (N,R&C) formulated in Montanide ISA 51 — 100 ug
  Other Names: Peptides (N, R & C) from P. vivax CS protein
  Arms: Group D
Other: Placebo — PLacebo: Isotonic saline solution
  Arms: Group E

SUMMARY:
This was a phase I double blind controlled vaccine trial, evaluating safety, tolerability and immunogenicity of mixtures of N, R and C LSP derived from the P. vivax CS protein formulated in two adjuvants Montanide ISA 720 and Montanide ISA 51.

The primary objective was to assess in malaria-naïve adults, the safety and reactogenicity of these peptides formulated in the two adjuvants

We recruited 40 healthy men and women volunteers from Cali, Colombia, a city non-endemic for malaria. Volunteers were 19--41 years of age and had no history of malaria. During a period of three months a total of 100 volunteers were assessed for eligibility criteria in order to select a total of 40 volunteers willing to participate in the clinical trial. By consecutive allocation, eight participants were allocated to each of the five experimental groups (A--E): four groups (A--D) were immunized with the vaccine formulations at two different dose concentrations and formulated in two different adjuvants. A control group (E) was injected with placebo (saline solution)

DETAILED DESCRIPTION:
The study corresponds to a clinical trial, randomized double-blind, controlled, dose escalation, Phase IB, which will assess the safety and immunogenicity of a mixture of synthetic peptides derived from CS protein of P. vivax, formulated in adjuvant Montanide ISA 720 and 51; in healthy men and nonpregnant women without previous history of malaria infection.

In order to optimize the vaccine dose, eligible participants were enrolled to receive three doses of vaccine containing peptide mixtures at a dose of 50 ug or 100 ug of each individual peptide, for a final dose of 150 ug or 300 ug respectively, in a volume of 0.5 mL. The previous clinical trial had indicated that doses between 30 ug and 100 ug produced better responses than lower doses. The first immunization dose (given at Month 0) contained the peptides N and C only, whereas the two boosting doses (given at Months 2 and 4) contained all three (N, R, and C) peptides (Table 1). Vaccination was performed by intramuscular injection in the deltoid muscle, alternating arms with each injection.

For safety reasons, participants assigned to the low vaccine dose groups were immunized first and only two weeks after initiation when no serious adverse events (SAE) had occurred, immunization of participants in the high-dose was started. Half of the participants assigned to receive placebo were immunized along with each dose level group. Clinical monitors and the IRBs of the University of Valle and IMC, evaluated the occurrence and severity of adverse events (AE) associated with immunization. The occurrence of more than three AE (severity grade 2 or higher) or one SAE related to the vaccine would have led to study termination. Participants who left the study were not replaced.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults (male and non-pregnant female) 18- 45 years old, without previously malaria infection (naïve volunteers), capable to pass a comprehension test on the study and able to provide written informed consent to participate in the trial.
* Use of adequate contraceptive method since the initiation of the study and until two months after the end of the study.
* No plans to travel to a malaria endemic area during the course of the study.
* Reachable by phone during the study period (1 year).
* No use of other vaccines since 3 months before the beginning of the study and during it.

Exclusion Criteria:

* Females who intend to become pregnant within the 3 months following the screening visit or who are pregnant at screening time, ascertained by urine or serum pregnancy test (B-HCG). Women who are breast-feeding will also be excluded. Reason for exclusion: The immunological changes accompanying pregnancy and lactation could alter the results of the assays performed. If a pathological condition appear, it could be carried to the vaccine.
* Duffy negative phenotype. Justification: Individuals with this phenotype are refractory to P. vivax infection.
* G-6-PD deficiency or any genetic defect (hemoglobinopathy). Justification: These conditions influence the development of P. vivax infection.
* History of previous experimental malaria vaccination. Justification: Individuals who have been previously immunized may show a response due to the past immunization and not to the present one.
* Clinical or laboratory evidence of significant systemic disease, including hepatic, renal, cardiac, immunologic or hematological disease.

Justification: The results of the study could have a negative impact on the study if volunteers are suffering from any of these diseases.

* Evidence of active hepatitis B or C or HIV infection. Justification: Serious underlying medical condition could affect the immunological responses of volunteers or could increase the risk or severity of adverse events associated with participation in this study.
* Clinically significant laboratory abnormalities as determined by the investigator(s).

Justification: Baseline abnormal laboratory values may indicate a serious underlying medical condition and also will make it difficult to evaluate AE´s during the conduct of the study.

• Known history of autoimmune (including inflammatory bowel disease, rheumatoid arthritis, lupus) or connective tissue disease.

Justification: Autoimmune diseases could affect the immunological responses of volunteers and could increase the risk to the volunteer.

• Individuals receiving treatment with steroids or non-steroidal anti-inflammatory drugs or any immunosuppressive therapy.

Justification: These drugs could affect the immunological responses of volunteers and could increase the risk to the volunteer.

* Known history of drug or alcohol abuse interfering with normal social function. Justification: Pharmaco-dependency alters the capacity of free decision and produce physical or psychiatric undesirable condition that could affect the study.
* Volunteers unable to give written informed consent or with difficulties to understand the study.

Justification: Volunteers must have the capacity to provide informed consent in order to participate in any research involving humans

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2005-07; Primary Completion 2006-03 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Safety and Immunogenicity of Plasmodium vivax CS Derived Long Synthetic Peptides Adjuvanted with Montanide ISA 720 or Montanide ISA 51 | 9 months

SECONDARY OUTCOMES:
Immunogenicity assessment | 9 month
  Specific anti CS antibodies determination (B cell response) and specific induction of IFNγ production (T cell response). All sera samples will be kept at -70° in Immunology Institute, FCVL or Asoclinic until use.
Adverse Events | 9 month
  Each AE will be written on CRF forms and will be immediately be informed to the clinical monitor and IRB. All volunteers will be followed until recovering it the initial condition. Additional physical examination and laboratory tests will be performed in case any relation between the AE and the immunogen needs to be established.
Safety Laboratories | 8 month
  Complete blood cell count, hepatic and renal function tests will be made on months 1, 2, 3, 6, 7 y 9 after the first immunization. Every change in the laboratory results will be reported on the corresponding CRF´s; severity associated with vaccination will be established. Specific studies will be made if it is necessary the AE end will be determined when these parameters will be normal.
B-cell response | 8 month
  Specific antibody titers will be measured by ELISA technique using the corresponding peptide (N, R, C) as coating antigen and the recognition of the native protein will be assessed by Immunofluorescence technique (IFAT) using P vivax sporozoites obtained by dissection of experimentally infected Anopheles mosquitoes [91] Antibody titers will be considered as positive at 1:100 dilution by ELISA and 1:40 by IFAT.
T-cell response evaluation | 8 month
  Cell mediated immune (CMI) responses will be evaluated will be made by the cytokines IFN-γ production using peripheral blood mononuclear cells (PBMC) using both ELIspot and ELISA techniques.
Cytokine Production Evaluation by ELISA | 8 month
  PBMC will be stimulated with each of the three peptides (N, R or C) in a concentration of 10ug/ml and cells cultures without the peptide will be used as negative control. PBMC stimulated with phyto-hemaglutinin (PHA) will be used as positive controls.
Cytokine Production by ELIspot | 8 month
  This evaluation will be made in two phases: First the cytokine production in total PBMC, which will be stimulated with CS protein derived peptides of different length. Second, positive samples for cytokine will be used to evaluate the production of cytokines by purified T lymphocytes subpopulations CD4+ or CD8+. This will determine the subpopulation responsible for cytokine production. A positive selection of cell subpopulations will be performed using anti-CD4+ / CD8+ coated pearls using MACS, and will be further used for ELIspot.

CONTACTS AND LOCATIONS:
Overall Officials: Myriam Arevalo-Herrera, PhD, Study Director — MVDC
Locations (2):
- Colombia (2):
  - Malaria Vaccine and Drug Testing Center, Cali, Valle del Cauca Department
  - Malaria Vaccine of Develepmente Center, Cali, Valle del Cauca Department

REFERENCES:
- [Background] Nussenzweig RS, Vanderberg J, Most H, Orton C. Protective immunity produced by the injection of x-irradiated sporozoites of plasmodium berghei. Nature. 1967 Oct 14;216(5111):160-2. doi: 10.1038/216160a0. No abstract available. PMID 6057225
- [Background] Clyde DF. Immunity to falciparum and vivax malaria induced by irradiated sporozoites: a review of the University of Maryland studies, 1971-75. Bull World Health Organ. 1990;68 Suppl(Suppl):9-12. PMID 2094597
- [Background] Herrington D, Davis J, Nardin E, Beier M, Cortese J, Eddy H, Losonsky G, Hollingdale M, Sztein M, Levine M, et al. Successful immunization of humans with irradiated malaria sporozoites: humoral and cellular responses of the protected individuals. Am J Trop Med Hyg. 1991 Nov;45(5):539-47. doi: 10.4269/ajtmh.1991.45.539. PMID 1951863
- [Background] Hoffman SL, Goh LM, Luke TC, Schneider I, Le TP, Doolan DL, Sacci J, de la Vega P, Dowler M, Paul C, Gordon DM, Stoute JA, Church LW, Sedegah M, Heppner DG, Ballou WR, Richie TL. Protection of humans against malaria by immunization with radiation-attenuated Plasmodium falciparum sporozoites. J Infect Dis. 2002 Apr 15;185(8):1155-64. doi: 10.1086/339409. Epub 2002 Apr 1. PMID 11930326
- [Background] Egan JE, Hoffman SL, Haynes JD, Sadoff JC, Schneider I, Grau GE, Hollingdale MR, Ballou WR, Gordon DM. Humoral immune responses in volunteers immunized with irradiated Plasmodium falciparum sporozoites. Am J Trop Med Hyg. 1993 Aug;49(2):166-73. doi: 10.4269/ajtmh.1993.49.166. PMID 8357078
- [Background] Romero P, Maryanski JL, Corradin G, Nussenzweig RS, Nussenzweig V, Zavala F. Cloned cytotoxic T cells recognize an epitope in the circumsporozoite protein and protect against malaria. Nature. 1989 Sep 28;341(6240):323-6. doi: 10.1038/341323a0. PMID 2477703
- [Background] Tsuji M, Romero P, Nussenzweig RS, Zavala F. CD4+ cytolytic T cell clone confers protection against murine malaria. J Exp Med. 1990 Nov 1;172(5):1353-7. doi: 10.1084/jem.172.5.1353. PMID 2146361
- [Background] Daubersies P, Thomas AW, Millet P, Brahimi K, Langermans JA, Ollomo B, BenMohamed L, Slierendregt B, Eling W, Van Belkum A, Dubreuil G, Meis JF, Guerin-Marchand C, Cayphas S, Cohen J, Gras-Masse H, Druilhe P. Protection against Plasmodium falciparum malaria in chimpanzees by immunization with the conserved pre-erythrocytic liver-stage antigen 3. Nat Med. 2000 Nov;6(11):1258-63. doi: 10.1038/81366. PMID 11062538
- [Background] Chappel JA, Rogers WO, Hoffman SL, Kang AS. Molecular dissection of the human antibody response to the structural repeat epitope of Plasmodium falciparum sporozoite from a protected donor. Malar J. 2004 Jul 29;3:28. doi: 10.1186/1475-2875-3-28. PMID 15283866
- [Background] Hoffman SL, Nussenzweig V, Sadoff JC, Nussenzweig RS. Progress toward malaria preerythrocytic vaccines. Science. 1991 Apr 26;252(5005):520-1. doi: 10.1126/science.2020852. No abstract available.
- [Background] Taylor-Robinson AW. Immunity to liver stage malaria: considerations for vaccine design. Immunol Res. 2003;27(1):53-70. doi: 10.1385/IR:27:1:53. PMID 12637768
- [Background] Cerami C, Frevert U, Sinnis P, Takacs B, Clavijo P, Santos MJ, Nussenzweig V. The basolateral domain of the hepatocyte plasma membrane bears receptors for the circumsporozoite protein of Plasmodium falciparum sporozoites. Cell. 1992 Sep 18;70(6):1021-33. doi: 10.1016/0092-8674(92)90251-7. PMID 1326407
- [Background] Frevert U, Sinnis P, Cerami C, Shreffler W, Takacs B, Nussenzweig V. Malaria circumsporozoite protein binds to heparan sulfate proteoglycans associated with the surface membrane of hepatocytes. J Exp Med. 1993 May 1;177(5):1287-98. doi: 10.1084/jem.177.5.1287. PMID 8478608
- [Background] Stoute JA, Slaoui M, Heppner DG, Momin P, Kester KE, Desmons P, Wellde BT, Garcon N, Krzych U, Marchand M. A preliminary evaluation of a recombinant circumsporozoite protein vaccine against Plasmodium falciparum malaria. RTS,S Malaria Vaccine Evaluation Group. N Engl J Med. 1997 Jan 9;336(2):86-91. doi: 10.1056/NEJM199701093360202. PMID 8988885
- [Background] Sun P, Schwenk R, White K, Stoute JA, Cohen J, Ballou WR, Voss G, Kester KE, Heppner DG, Krzych U. Protective immunity induced with malaria vaccine, RTS,S, is linked to Plasmodium falciparum circumsporozoite protein-specific CD4+ and CD8+ T cells producing IFN-gamma. J Immunol. 2003 Dec 15;171(12):6961-7. doi: 10.4049/jimmunol.171.12.6961. PMID 14662904
- [Background] Kester KE, McKinney DA, Tornieporth N, Ockenhouse CF, Heppner DG Jr, Hall T, Wellde BT, White K, Sun P, Schwenk R, Krzych U, Delchambre M, Voss G, Dubois MC, Gasser RA Jr, Dowler MG, O'Brien M, Wittes J, Wirtz R, Cohen J, Ballou WR; RTS,S Malaria Vaccine Evaluation Group. A phase I/IIa safety, immunogenicity, and efficacy bridging randomized study of a two-dose regimen of liquid and lyophilized formulations of the candidate malaria vaccine RTS,S/AS02A in malaria-naive adults. Vaccine. 2007 Jul 20;25(29):5359-66. doi: 10.1016/j.vaccine.2007.05.005. Epub 2007 May 30. PMID 17574311
- [Background] Kester KE, Cummings JF, Ockenhouse CF, Nielsen R, Hall BT, Gordon DM, Schwenk RJ, Krzych U, Holland CA, Richmond G, Dowler MG, Williams J, Wirtz RA, Tornieporth N, Vigneron L, Delchambre M, Demoitie MA, Ballou WR, Cohen J, Heppner DG Jr; RTS,S Malaria Vaccine Evaluation Group. Phase 2a trial of 0, 1, and 3 month and 0, 7, and 28 day immunization schedules of malaria vaccine RTS,S/AS02 in malaria-naive adults at the Walter Reed Army Institute of Research. Vaccine. 2008 Apr 24;26(18):2191-202. doi: 10.1016/j.vaccine.2008.02.048. Epub 2008 Mar 13. PMID 18387719
- [Background] Bojang KA, Milligan PJ, Pinder M, Vigneron L, Alloueche A, Kester KE, Ballou WR, Conway DJ, Reece WH, Gothard P, Yamuah L, Delchambre M, Voss G, Greenwood BM, Hill A, McAdam KP, Tornieporth N, Cohen JD, Doherty T; RTS, S Malaria Vaccine Trial Team. Efficacy of RTS,S/AS02 malaria vaccine against Plasmodium falciparum infection in semi-immune adult men in The Gambia: a randomised trial. Lancet. 2001 Dec 8;358(9297):1927-34. doi: 10.1016/S0140-6736(01)06957-4. PMID 11747915
- [Background] Alonso PL, Sacarlal J, Aponte JJ, Leach A, Macete E, Milman J, Mandomando I, Spiessens B, Guinovart C, Espasa M, Bassat Q, Aide P, Ofori-Anyinam O, Navia MM, Corachan S, Ceuppens M, Dubois MC, Demoitie MA, Dubovsky F, Menendez C, Tornieporth N, Ballou WR, Thompson R, Cohen J. Efficacy of the RTS,S/AS02A vaccine against Plasmodium falciparum infection and disease in young African children: randomised controlled trial. Lancet. 2004 Oct 16-22;364(9443):1411-20. doi: 10.1016/S0140-6736(04)17223-1. PMID 15488216
- [Background] Bejon P, Lusingu J, Olotu A, Leach A, Lievens M, Vekemans J, Mshamu S, Lang T, Gould J, Dubois MC, Demoitie MA, Stallaert JF, Vansadia P, Carter T, Njuguna P, Awuondo KO, Malabeja A, Abdul O, Gesase S, Mturi N, Drakeley CJ, Savarese B, Villafana T, Ballou WR, Cohen J, Riley EM, Lemnge MM, Marsh K, von Seidlein L. Efficacy of RTS,S/AS01E vaccine against malaria in children 5 to 17 months of age. N Engl J Med. 2008 Dec 11;359(24):2521-32. doi: 10.1056/NEJMoa0807381. Epub 2008 Dec 8. PMID 19064627
- [Background] Abdulla S, Oberholzer R, Juma O, Kubhoja S, Machera F, Membi C, Omari S, Urassa A, Mshinda H, Jumanne A, Salim N, Shomari M, Aebi T, Schellenberg DM, Carter T, Villafana T, Demoitie MA, Dubois MC, Leach A, Lievens M, Vekemans J, Cohen J, Ballou WR, Tanner M. Safety and immunogenicity of RTS,S/AS02D malaria vaccine in infants. N Engl J Med. 2008 Dec 11;359(24):2533-44. doi: 10.1056/NEJMoa0807773. Epub 2008 Dec 8. PMID 19064623
- [Background] Herrera S, Bonelo A, Perlaza BL, Valencia AZ, Cifuentes C, Hurtado S, Quintero G, Lopez JA, Corradin G, Arevalo-Herrera M. Use of long synthetic peptides to study the antigenicity and immunogenicity of the Plasmodium vivax circumsporozoite protein. Int J Parasitol. 2004 Dec;34(13-14):1535-46. doi: 10.1016/j.ijpara.2004.10.009. PMID 15582530
- [Background] Herrera S, Perlaza BL, Bonelo A, Arevalo-Herrera M. Aotus monkeys: their great value for anti-malaria vaccines and drug testing. Int J Parasitol. 2002 Dec 4;32(13):1625-35. doi: 10.1016/s0020-7519(02)00191-1. PMID 12435447
- [Background] Herrera S, Bonelo A, Perlaza BL, Fernandez OL, Victoria L, Lenis AM, Soto L, Hurtado H, Acuna LM, Velez JD, Palacios R, Chen-Mok M, Corradin G, Arevalo-Herrera M. Safety and elicitation of humoral and cellular responses in colombian malaria-naive volunteers by a Plasmodium vivax circumsporozoite protein-derived synthetic vaccine. Am J Trop Med Hyg. 2005 Nov;73(5 Suppl):3-9. doi: 10.4269/ajtmh.2005.73.3. PMID 16291760
- [Background] Pye D, Vandenberg KL, Dyer SL, Irving DO, Goss NH, Woodrow GC, Saul A, Alving CR, Richards RL, Ballou WR, Wu MJ, Skoff K, Anders RF. Selection of an adjuvant for vaccination with the malaria antigen, MSA-2. Vaccine. 1997 Jun;15(9):1017-23. doi: 10.1016/s0264-410x(96)00289-7. PMID 9261951
- [Background] Peters BS, Jaoko W, Vardas E, Panayotakopoulos G, Fast P, Schmidt C, Gilmour J, Bogoshi M, Omosa-Manyonyi G, Dally L, Klavinskis L, Farah B, Tarragona T, Bart PA, Robinson A, Pieterse C, Stevens W, Thomas R, Barin B, McMichael AJ, McIntyre JA, Pantaleo G, Hanke T, Bwayo J. Studies of a prophylactic HIV-1 vaccine candidate based on modified vaccinia virus Ankara (MVA) with and without DNA priming: effects of dosage and route on safety and immunogenicity. Vaccine. 2007 Mar 1;25(11):2120-7. doi: 10.1016/j.vaccine.2006.11.016. Epub 2006 Nov 27. PMID 17250931
- [Background] Aucouturier J, Ascarateil S, Dupuis L. The use of oil adjuvants in therapeutic vaccines. Vaccine. 2006 Apr 12;24 Suppl 2:S2-44-5. doi: 10.1016/j.vaccine.2005.01.116. PMID 16823921
- [Background] O'Hagan DT, Valiante NM. Recent advances in the discovery and delivery of vaccine adjuvants. Nat Rev Drug Discov. 2003 Sep;2(9):727-35. doi: 10.1038/nrd1176. PMID 12951579
- [Background] Arevalo-Herrera M, Solarte Y, Yasnot MF, Castellanos A, Rincon A, Saul A, Mu J, Long C, Miller L, Herrera S. Induction of transmission-blocking immunity in Aotus monkeys by vaccination with a Plasmodium vivax clinical grade PVS25 recombinant protein. Am J Trop Med Hyg. 2005 Nov;73(5 Suppl):32-7. doi: 10.4269/ajtmh.2005.73.32. PMID 16291764
- [Background] Arevalo-Herrera M, Castellanos A, Yazdani SS, Shakri AR, Chitnis CE, Dominik R, Herrera S. Immunogenicity and protective efficacy of recombinant vaccine based on the receptor-binding domain of the Plasmodium vivax Duffy binding protein in Aotus monkeys. Am J Trop Med Hyg. 2005 Nov;73(5 Suppl):25-31. doi: 10.4269/ajtmh.2005.73.5_suppl.0730025. PMID 16291763
- [Background] Valderrama-Aguirre A, Quintero G, Gomez A, Castellanos A, Perez Y, Mendez F, Arevalo-Herrera M, Herrera S. Antigenicity, immunogenicity, and protective efficacy of Plasmodium vivax MSP1 PV200l: a potential malaria vaccine subunit. Am J Trop Med Hyg. 2005 Nov;73(5 Suppl):16-24. doi: 10.4269/ajtmh.2005.73.16. PMID 16291762
- [Background] Bell BA, Wood JF, Bansal R, Ragab H, Cargo J 3rd, Washington MA, Wood CL, Ware LA, Ockenhouse CF, Yadava A. Process development for the production of an E. coli produced clinical grade recombinant malaria vaccine for Plasmodium vivax. Vaccine. 2009 Feb 25;27(9):1448-53. doi: 10.1016/j.vaccine.2008.12.027. Epub 2009 Jan 10. PMID 19138714
- [Background] Hu J, Chen Z, Gu J, Wan M, Shen Q, Kieny MP, He J, Li Z, Zhang Q, Reed ZH, Zhu Y, Li W, Cao Y, Qu L, Cao Z, Wang Q, Liu H, Pan X, Huang X, Zhang D, Xue X, Pan W. Safety and immunogenicity of a malaria vaccine, Plasmodium falciparum AMA-1/MSP-1 chimeric protein formulated in montanide ISA 720 in healthy adults. PLoS One. 2008 Apr 9;3(4):e1952. doi: 10.1371/journal.pone.0001952. PMID 18398475
- [Background] Malkin E, Hu J, Li Z, Chen Z, Bi X, Reed Z, Dubovsky F, Liu J, Wang Q, Pan X, Chen T, Giersing B, Xu Y, Kang X, Gu J, Shen Q, Tucker K, Tierney E, Pan W, Long C, Cao Z. A phase 1 trial of PfCP2.9: an AMA1/MSP1 chimeric recombinant protein vaccine for Plasmodium falciparum malaria. Vaccine. 2008 Dec 9;26(52):6864-73. doi: 10.1016/j.vaccine.2008.09.081. Epub 2008 Oct 16. PMID 18930094
- [Background] Wu Y, Ellis RD, Shaffer D, Fontes E, Malkin EM, Mahanty S, Fay MP, Narum D, Rausch K, Miles AP, Aebig J, Orcutt A, Muratova O, Song G, Lambert L, Zhu D, Miura K, Long C, Saul A, Miller LH, Durbin AP. Phase 1 trial of malaria transmission blocking vaccine candidates Pfs25 and Pvs25 formulated with montanide ISA 51. PLoS One. 2008 Jul 9;3(7):e2636. doi: 10.1371/journal.pone.0002636. PMID 18612426
- [Background] Roestenberg M, Remarque E, de Jonge E, Hermsen R, Blythman H, Leroy O, Imoukhuede E, Jepsen S, Ofori-Anyinam O, Faber B, Kocken CH, Arnold M, Walraven V, Teelen K, Roeffen W, de Mast Q, Ballou WR, Cohen J, Dubois MC, Ascarateil S, van der Ven A, Thomas A, Sauerwein R. Safety and immunogenicity of a recombinant Plasmodium falciparum AMA1 malaria vaccine adjuvanted with Alhydrogel, Montanide ISA 720 or AS02. PLoS One. 2008;3(12):e3960. doi: 10.1371/journal.pone.0003960. Epub 2008 Dec 18. PMID 19093004
- See also: Related Info — http://www.inmuno.org